CLINICAL TRIAL: NCT04691557
Title: Evaluation of the Effectiveness of User-focused Mobile Health Application on Asthma Control and Self-efficacy in Adolescents With Asthma: a Randomized Controlled Trial Protocol
Brief Title: Mobile Health Application for Adolescents With Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Nimet KARATAS, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2012KAEK20
Record Dates: First submitted 2020-12-23; First posted 2020-12-31 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Adolescent; Nursing Care; Asthma in Children; Self Efficacy
Keywords: Asthma Control; Nursing care; Mobile Health; Self-Efficacy; Randomized Controlled Trial; Adolescent

STUDY DESIGN:
Intervention Model Description: A self-efficacy theory based, randomized, 4-week, parallel group study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group receives the YoungAsthma developing for the smartphone or tablet additionally usual nursing care.
  Interventions: Other: Mobile Health Application
- Control Group (Active Comparator): The control group receives the usual nursing care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Mobile Health Application — YoungAsthma is a web-based mobile health app has been developing user-focused for adolescents with asthma and evidence-based by the research team. It is the integrated version of the knowledge content to software that enables effective management of asthma by strengthening the interaction between adolescents and healthcare professionals.
  Arms: Intervention Group
Other: Usual Care — Adolescents in the control group, an asthma training covering also individualized specific conditions is provided by specialist training nurse for 15-30 minutes in the nursing room of the outpatient clinic for all children. In this nursing intervention that is only one-off and consist face-to-face training with adolescents video and visual materials included in the routine of the outpatient clinic for the use of devices and drugs are used.
  Arms: Control Group

SUMMARY:
Mobile health applications (mHealth apps) are an opportunity offered by developing technology which in widely used among youths. The evidence regarding mHealth apps suggests that the apps can be safer and more feasible if are developed by healthcare team. Healthcare professionals have a major role to play in developing mHealth apps of good interventions.

DETAILED DESCRIPTION:
This study aims at developing the mHealth application (YoungAsthma) and evaluating the effectiveness of YoungAsthma app on the mean score of the asthma control test and self-efficacy scale in adolescents with asthma. This study is a self-efficacy theory-based, 4-week, randomized parallel group study. Participants will be randomized to either the intervention or control group in a 1:1 ratio. Adolescents will be randomly allocated to intervention (YoungAsthma which is a user-focused mHealth app) or control group (Usual care). The study protocol is conducted in accord with the Standard Protocol Items: Recommendations for Interventional Trials (SPIRIT 2013 Statement) (Chan et al., 2013), the RCT is perform by the Consolidated Standards of Reporting Trials (CONSORT) (Moher et al., 2010) and the mHealth app is identified according to the mERA guideline (Agarwal et al., 2016).

ELIGIBILITY:
Inclusion Criteria:

* Having ability to speak, read and write Turkish at a sufficient level,
* Having a diagnosis of asthma for at least a year,
* Having an asthma control test score of 19 or below,
* Having ability to use mobile devices,
* Having a mobile device with an internet connection to login to the mHealth App.

Exclusion Criteria:

* Having an internet access problem,
* Having a psychiatric medical diagnosis

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Self-Efficacy | Assessment of change of the self-efficacy from baseline to 4 weeks will be done.
  Self-efficacy will be evaluated by Asthmatic Child and Adolescent Self-Efficacy Scale (ACASES) (Schlösser & Havermans, 1992).
Asthma Control | Assessment of change of the asthma control from baseline to 4 weeks will be done.
  Asthma control will be evaluated by the Asthma Control Test (ACT) (Liu et al., 2007).

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul ISLER DALGIC, Professor, Study Director — Akdeniz University; Aysen BINGOL, Professor, Study Chair — Akdeniz University
Locations (2):
- Turkey (Türkiye) (2):
  - Akdeniz University Hospital, Antalya, None Selected
  - Antalya Education and Research Hospital, Antalya, None Selected

IPD SHARING:
Plan to Share IPD: No
It has not been yet decided. After the study is finalized, the plan to share individual participant data will be done.

REFERENCES:
- [Derived] Karatas N, Isler A, Bingol A. Enhancing Adolescent Asthma Control and Self-Efficacy: A Decision Tree Analysis of a Mobile Health Application in a Randomized Controlled Trial. J Eval Clin Pract. 2025 Sep;31(6):e70266. doi: 10.1111/jep.70266. PMID 40928010